CLINICAL TRIAL: NCT06955780
Title: Examining the Effect of the Emotional Freedom Techniques on Burnout in Rehabilitation Therapists
Brief Title: Emotional Freedom Techniques on Burnout in Therapists
Acronym: EFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Indianapolis (Other)
Responsible Party: Principal Investigator, Erin Peterson DHSc, Assistant Professor of Practice, University of Indianapolis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01870
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Burnout; Anxiety; Distress, Emotional
Keywords: burnout; emotional freedom techniques; EFT; occupational therapy; distress
MeSH Terms: conditions — Burnout, Psychological; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Emotional Freedom Techniques — Emotional Freedom Techniques

SUMMARY:
The goal of this study is to investigate the effectiveness of Emotional Freedome Techniques (EFT) on burnout in rehabilitation therapists. The main question[s] it aims to answer [is/are]:

1. Does a single session of EFT reduce burnout in therapists immediately and/or one month later as measured by the short version of the Burnout Assessment Tool (BAT-S)?
2. Does a single session of EFT reduce Subjective Units of Distress (SUDS) data related to burnout in therapists immediately and/or one month later?
3. Do clinicians with more years of experience have overall lower levels of burnout as measured by the BAT-S?
4. Are there significant differences in the level of burnout amongst occupational or physical therapists?

Participants will:

* Complete the demographic survey using the Qualtrics link. Information pertaining to age, gender, years of work experience, professional discipline, workplace setting, etc. will be gathered.
* Complete a short 12-item questionnaire (Burnout Assessment Tool - Short [BAT-S]) that immediately follows the demographic questions. Questions will be related to experiencing feelings of burnout.
* Attend a free, live, virtual wellness session. Before the session begins, you will be asked to privately answer three questions related to current levels of work distress, despair, and anxiety using a Qualtrics link. During the wellness session, the research team consisting of the PI and student researchers will describe what Emotional Freedom Techniques (EFT) is and how it is performed. The research team will then lead participants through EFT with you performing the technique on yourself.
* Immediately following the session, you will be asked to privately answer the three questions relating to work distress, despair, and anxiety again using a Qualtrics link.
* One month after completing the session, you will receive an email containing a Qualtrics link to answer the work distress, despair, and anxiety questions again, as well as the BAT-S in order for the researchers to collect follow-up data.

DETAILED DESCRIPTION:
Healthcare employees experience various difficulties, and burnout is one of the most pressing issues in the field (Bridgeman et al., 2018; Knox et al., 2018). Emotional Freedom Techniques (EFT), commonly called "tapping," is an emerging psychophysiological intervention that combines elements from cognitive therapy, exposure therapy, and acupressure (Church, 2019; Church et al., 2022). The purpose of this study is to investigate the effectiveness of EFT on burnout in rehabilitation therapists. Participants will be members of the American Society of Hand Therapists (ASHT) who are actively employed as occupational therapy or physical therapy practitioners. To recruit participants, researchers will complete the ASHT research division's application for participant recruitment. If the application is denied, researchers will recruit participants through social media. Participants will attend a free, one-hour live virtual wellness session held on a virtual meeting platform. If they choose to participate in the study, they will be directed to a Qualtrics survey to complete the informed consent, demographics, and the Burnout Assessment Tool. During the session, the researchers will guide participants through EFT, collecting Subjective Units of Distress Scale (SUDS) and expanded SUDS data immediately prior to and following the intervention. Additionally, researchers will collect follow-up data using the BAT-S, SUDS, and expanded SUDS questions one month later. Researchers will perform descriptive statistics to analyze demographic data and use SPSS with appropriate statistical tests to explore relationships between the BAT-S, SUDS, and expanded SUDS data from the pre, post, and follow-up data.

ELIGIBILITY:
Inclusion Criteria: (a) the ability to read and speak English, (b) 18 years of age or older, and (c) actively working in direct patient care.

Exclusion Criteria:

* Exclusion criteria consisted of individuals who were not practicing therapists, such as managers, therapy aides, or technicians. Following initial recruitment efforts, the researchers were invited to conduct the virtual EFT session for therapy employees of a private practice. Due to this, the researchers expanded the inclusion criteria to include speech therapists employed at this facility. All other inclusion and exclusion criteria remained the same.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-10-22 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
Subjective Units of Distress | before, immediately after, and at the one-month follow-up of the EFT session
  The SUDS is a rating scale used with EFT to measure individuals' current subjective units of distress. The scale ranges from 0 to 10, with 0 being no distress and 10 being the highest level of distress (Church, 2019).
Burnout Assessment Tool (BAT) | before EFT session and at the one-month follow-up
  The BAT is a self-report, Likert-scale questionnaire used to measure burnout. The developers divided burnout into four core scales: exhaustion, mental distance, cognitive impairment, and emotional impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Indianapolis, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol, ICF
Time Frame: Start date (now) until 1/1/2032
Access Criteria: Upon request

REFERENCES:
- [Background] Church D, Stapleton P, Vasudevan A, O'Keefe T. Clinical EFT as an evidence-based practice for the treatment of psychological and physiological conditions: A systematic review. Front Psychol. 2022 Nov 10;13:951451. doi: 10.3389/fpsyg.2022.951451. eCollection 2022. PMID 36438382
- [Background] Church, D. (2019). The EFT Manual (4th ed.) Energy Psychology Press.